CLINICAL TRIAL: NCT03062657
Title: An Investigation of the Metal Concentration in Patients Implanted With the PRESTIGE LP™ Cervical Disc at Two Contiguous Levels in the Cervical Spine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prematurely as agreed by the FDA. The FDA were satisfied that no further data was required, despite the total number of patients who completed the study in full not being the agreed upon number.
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD1701
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cervical Degenerative Disc Disease; Radiculopathy; Myelopathy
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PRESTIGE LP (Experimental): Patients receive surgical treatment with the PRESTIGE LP™ Cervical Disc at two contiguous cervical levels from C3-C7.
  Interventions: Device: PRESTIGE LP™ Cervical Disc

INTERVENTIONS:
Device: PRESTIGE LP™ Cervical Disc — The PRESTIGE LP™ Cervical Disc is an artificial cervical disc comprising of two low-profile metal plates that interface through a ball and trough mechanism, permitting segmental spinal motion. The PRESTIGE LP™ Cervical Disc was approved by the Food and Drug Administration (FDA) to be used at a single and two contiguous levels.

SUMMARY:
This clinical study will assess the metal concentrations present in the blood serum of patients who receive surgical treatment with the PRESTIGE LP™ Cervical Disc at two contiguous cervical levels from C3-C7. The information obtained from this clinical investigation will be used to support the post market surveillance for a PMA supplement for the PRESTIGE LP™ Cervical Disc implanted at two contiguous levels.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to participate in this study:

1. Has cervical degenerative disc disease at two (2) contiguous cervical levels (from C3 to C7) requiring surgical treatment and involving intractable radiculopathy, myelopathy or both;
2. Has a herniated disc and/or osteophyte formation at each level to be treated that is producing symptomatic nerve root and/or spinal cord compression. The condition is documented by patient history (e.g., neck and/or arm pain, functional deficit and /or neurological deficit), and the requirement for surgical treatment is evidenced by radiographic studies (e.g., CT, MRI, x-rays, etc.);
3. Has been unresponsive to non-operative treatment for at least six weeks or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of continued non-operative therapy;
4. Has no previous surgical intervention at the involved levels or any other planned/staged surgical procedure at the involved levels;
5. Has preoperative neck pain score ≥ 8 based on the preoperative Neck and Arm Pain Questionnaire;
6. Must be at least 18 years of age and be skeletally mature at the time of surgery;
7. If a female of childbearing potential, patient is non-pregnant, non-nursing, and agrees not to become pregnant during the study period;
8. Is willing to comply with the study plan and sign the Patient Informed Consent Form.

Exclusion Criteria:

A patient will be excluded from participating in this study for any of the following reasons:

1. Has a cervical spine condition other than symptomatic cervical degenerative disease requiring surgical treatment at the involved levels;
2. Has documented or diagnosed cervical instability relative to contiguous segments at either level, defined by dynamic (flexion/extension) radiographs showing:

   1. Sagittal plane translation > 3.5 mm, or
   2. Sagittal plane angulation > 20°
3. Has more than two cervical levels requiring surgical treatment;
4. Has severe pathology of the facet joints of the involved vertebral bodies;
5. Has had previous surgical intervention at either one or both of the involved levels;
6. Has been previously diagnosed with osteopenia or osteomalacia;
7. Has any of the following that may be associated with a diagnosis of osteoporosis (If "Yes" to any of the below risk factors, a DEXA Scan will be required to determine eligibility.):

   1. . Postmenopausal non-Black female over 60 years of age who weighs less than 140 pounds.
   2. Postmenopausal female who has sustained a non-traumatic hip, spine or wrist fracture.
   3. Male over the age of 70.
   4. Male over the age of 60 who has sustained a non-traumatic hip or spine fracture.

   If the level of BMD is a T score of -3.5 or lower (i.e., -3.6, -3.7, etc.) or a T score of -2.5 or lower (i.e., -2.6, -2.7 etc.) with vertebral crush fracture, then the patient is excluded from the study
8. Has presence of spinal metastases;
9. Has overt or active bacterial infection, either local or systemic;
10. Has chronic or acute renal failure or prior history of renal disease;
11. Has a documented allergy or intolerance to titanium, or a titanium alloy;
12. Is mentally incompetent. (If questionable, obtain psychiatric consult);
13. Is a prisoner;
14. Is pregnant;
15. Has received drugs that may interfere with bone metabolism within two weeks prior to the planned date of spinal surgery (e.g., steroids or methotrexate), excluding routine perioperative anti-inflammatory drugs;
16. Has history of an endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's Disease, renal osteodystrophy, Ehlers-Danlos Syndrome, or osteogenesis imperfecta);
17. Has a condition that requires postoperative medications that interfere with the stability of the implant, such as steroids. (This does not include low-dose aspirin for prophylactic anticoagulation and routine perioperative anti-inflammatory drugs.);
18. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following implantation.
19. Is currently taking or has had chronic usage of certain prescription medications (e.g., Cloxacillin, an antibiotic used for prophylaxis against surgical infections, and/or Clotrimazole).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Todd H. Lanman, M.D., INC., Beverly Hills, California
  - Beaumont Hospital, Royal Oak, Michigan
  - Kellogg M.D., Brain & Spine, Portland, Oregon
  - Lexington Brain and Spine, West Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRESTIGE LP
Started | 25
6 Week Follow-Up | 25
3 Month Follow-Up | 18
6 Month Follow-Up | 17
Completed | 19
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Titanium, Vanadium, and Aluminum in the Blood Serum
Description: The concentrations of Titanium, Vanadium, and Aluminum at different time points will be summarized using mean and standard deviation.
  One participant did not receive metal concentration analysis at baseline, therefore the baseline number of participants for these measures N = 24.
Time Frame: Preoperative, 6 weeks, and 12 months
Population: Due to patient drop out not all patients attended every visit
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 24
ng/ml
  Titanium at Preoperative | 0.2253 (0.2264)
  Titanium at 6 weeks: number analyzed (Participants) | 21
  Titanium at 6 weeks | 2.7268 (1.4223)
  Titanium at 12 months: number analyzed (Participants) | 18
  Titanium at 12 months | 4.8485 (2.6315)
  Vanadium at Preoperative | 0.0522 (0.1676)
  Vanadium at 6 weeks: number analyzed (Participants) | 21
  Vanadium at 6 weeks | 0.0508 (0.0371)
  Vanadium at 12 months: number analyzed (Participants) | 18
  Vanadium at 12 months | 0.0538 (0.0222)
  Aluminum at Preoperative | 1.1 (1.1)
  Aluminum at 6 weeks: number analyzed (Participants) | 20
  Aluminum at 6 weeks | 1.3 (1.6)
  Aluminum at 12 months: number analyzed (Participants) | 18
  Aluminum at 12 months | 1.0 (0.7)

2. Secondary Outcome: Number of Participants Who Achieved Overall Success
Description: The patients enrolled in the study who receive the PRESTIGE LP™ Cervical Disc at two contiguous levels will be considered an overall success if the following criteria are met:
  1. NDI score improvement of at least 15 points from baseline;
  2. Maintenance or improvement in neurological status;
  3. No serious AE classified as implant associated/related or implant/surgical procedure associated/related;
  4. No secondary surgical procedure classified as a "failure".
Time Frame: 3, 6, and 12 months
Population: 17 patients data are presented at 3 months 16 patients data are presented at 6 months 18 patients data are presented at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 18
Participants
  3 months: number analyzed (Participants) | 17
  3 months: Overall Success Achieved | 12
  3 months: Overall Success Not Achieved | 5
  6 months: number analyzed (Participants) | 16
  6 months: Overall Success Achieved | 11
  6 months: Overall Success Not Achieved | 5
  12 months: Overall Success Achieved | 12
  12 months: Overall Success Not Achieved | 6

3. Secondary Outcome: Number of Participants Who Achieved NDI Success
Description: The self-administered Neck Disability Index (NDI) Questionnaire will be used. Success for each individual patient will be defined as pain/disability improvement postoperatively according to the following definition:
  Preoperative Score - Postoperative Score > 15
Time Frame: 3, 6, and 12 months
Population: Due to drop out, not all patients were present for each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 19
Participants
  3 Months: number analyzed (Participants) | 18
  3 Months: NDI Success Achieved | 13
  3 Months: NDI Success Not Achieved | 5
  6 Months: number analyzed (Participants) | 17
  6 Months: NDI Success Achieved | 12
  6 Months: NDI Success Not Achieved | 5
  12 Months: NDI Success Achieved | 14
  12 Months: NDI Success Not Achieved | 5

4. Secondary Outcome: Neck Pain and Arm Pain
Description: Numerical rating scales adapted in part from Measuring Health (McDowell and Newell, 1996) will be used to evaluate neck pain and arm pain.
  Intensity of pain is ranked from 0-10 with 0 being no pain and 10 being pain as bad as it could be; duration of pain is ranked from 0-10 with 0 being none of the time and 10 being pain all of the time.
  The pain score is derived by adding the numerical rating scores from the pain intensity and duration scales. Therefore the total pain is ranked between 0-20 with 0 being no pain, none of the time; and 20 being maximum pain, constantly.
Time Frame: Preoperative, 3, 6, and 12 months
Population: Due to drop out, not all patients were present for each visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 25
Score on a scale
  Neck Pain at Preoperative | 14.4 (3.0)
  Neck Pain at 3 Months: number analyzed (Participants) | 18
  Neck Pain at 3 Months | 6.2 (5.8)
  Neck Pain at 6 Months: number analyzed (Participants) | 17
  Neck Pain at 6 Months | 7.7 (5.8)
  Neck Pain at 12 Months: number analyzed (Participants) | 19
  Neck Pain at 12 Months | 8.1 (5.7)
  Arm Pain at Preoperative | 11.9 (4.9)
  Arm Pain at 3 Months: number analyzed (Participants) | 18
  Arm Pain at 3 Months | 4.8 (6.4)
  Arm Pain at 6 Months: number analyzed (Participants) | 17
  Arm Pain at 6 Months | 5.4 (6.4)
  Arm Pain at 12 Months: number analyzed (Participants) | 19
  Arm Pain at 12 Months | 5.1 (6.5)

5. Secondary Outcome: Number of Participants Who Achieved Neurological Success
Description: Neurological status is based on motor function, sensory function, and reflexes. Each of the categories is comprised of a number of elements. Postoperative evaluations of each element will be compared to the preoperative evaluations. Success will be defined as maintenance or improvement in each element for the time period evaluated.
Time Frame: 3, 6, and 12 months
Population: Due to drop out, not all patients were present for each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 18
Participants
  3 Months: number analyzed (Participants) | 17
  3 Months: Overall Neurological Success Achieved | 16
  3 Months: Overall Neurological Success Not Achieved | 1
  6 Months: number analyzed (Participants) | 14
  6 Months: Overall Neurological Success Achieved | 14
  6 Months: Overall Neurological Success Not Achieved | 0
  12 Months: Overall Neurological Success Achieved | 15
  12 Months: Overall Neurological Success Not Achieved | 3

6. Secondary Outcome: Number of Participants Who Underwent Secondary Surgery at Index Level
Description: Some AEs or treatment failures may lead to a secondary surgical intervention at an operated index level. All patients undergoing a secondary surgical intervention at any operated index level will be followed.
Time Frame: 3, 6, and 12 months
Population: Due to participant drop-out/missed visits, the number of participants per timepoint varies.
Measure: Count of Participants; unit: Participants
Arm/Group | PRESTIGE LP
Number analyzed (Participants) | 25
Participants
  3 Months | 0
  6 Months: number analyzed (Participants) | 17
  6 Months | 0
  12 Months: number analyzed (Participants) | 19
  12 Months | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to participant completion; specifically the pre-operative, 6 weeks, 3-months, 6-months and 12-months follow-up visits.
Arm/Group | PRESTIGE LP
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRESTIGE LP (N=25)
Arm Pain (Non-Cervical) (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Cord Disturbance (Nervous system disorders) | 1 (1)
Other Pain (General disorders) | 2 (2)
Spinal Event (Cervical Non-Study Surgery) (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRESTIGE LP (N=25)
Dysphagia/Dysphonia (Grade 1/2) (Gastrointestinal disorders) | 2 (3)
Neck and/or Arm Pain (Grade 1/2) (Musculoskeletal and connective tissue disorders) | 6 (9)
Neurological (Grade 1/2) (Nervous system disorders) | 7 (11)
Other Pain (Grade 1/2) (General disorders) | 5 (9)
Trauma (Grade 1/2) (Injury, poisoning and procedural complications) | 2 (2)

LIMITATIONS AND CAVEATS:
In agreement with the FDA, the study was terminated early, this lead to a sample size smaller than initially planned (30 planned, 25 enrolled). A short sample period was also used, however this was in agreement with the FDA based on previous evidence that the sample period would be sufficient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03062657/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT03062657/SAP_001.pdf